CLINICAL TRIAL: NCT03660280
Title: Probiotics to Treat "Inflammatory Depression" - a Randomized Controlled Trial
Brief Title: Probiotics to Treat "Inflammatory Depression"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Daniel Lindqvist, MD, PhD, Ass Prof, Region Skane
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018/379
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Depression
Keywords: Inflammation
MeSH Terms: conditions — Depression; Inflammation | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Intervention will be add-on specific probiotic to ongoing treatment with antidepressant medication or Cognitive Behavioral Therapy (CBT). Subjects will be randomized to placebo or probiotic. To assure a balanced subject recruitment, block randomization within strata (ongoing treatment with CBT, antidepressant or both) will be performed. Blood sampling and symptom rating scales will be completed at baseline, at weeks 4 and 8 (end of study). Feces will be collected at baseline and end of study. Biomarkers (from baseline, week 4 and week 8) will be analyzed after the study. Subjects will be recruited from outpatient or inpatient settings, Psychiatry Skåne or primary care clinics in Skåne, Sweden. Subjects will be recruited via clinical referrals, but also via ads.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental)
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Specific probiotic lactobacilli (added to stabilized ongoing treatment)
  Arms: Probiotics
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The main aims of this project are to test if: i) Specific probiotic lactobacilli (added to stabilized ongoing treatment) are efficacious in treating depressive symptoms in individuals with low-grade inflammation, defined using high sensitivity C-reactive protein (hs-CRP) and BMI. ii) This effect is mediated through decrease of inflammation, estimated by treatment-associated changes in blood and faeces biomarkers. Secondary aims are to investigate the relationship between specific depressive symptoms and inflammation and if there is a correlation between certain pro-inflammatory or metabolic markers and depression.

ELIGIBILITY:
Inclusion Criteria:

1. Age, 18-85
2. Depressive episode according to the DSM-V
3. MADRS-M score >18
4. All subjects will be stable on an antidepressant medication or in Cognitive Behavioural Therapy (CBT) for >4 weeks
5. Subjects will be willing not to significantly alter their diet during the period of the study
6. A hs-CRP value ≥1mg/L and BMI >25

Exclusion Criteria:

1. Serious or unstable medical illness that in the investigator's opinion could compromise response to treatment or interpretation of study results.
2. Known or suspected allergy to the study compounds.
3. Ongoing infection.
4. A diagnosis of psychotic disorder, bipolar disorder, personality disorder mental retardation, dementia, or individual whom, due to other causes, lack the ability to make an informed decision.
5. Ongoing ECT.
6. Patients who, in the investigator's judgment, pose a current, serious suicidal.
7. A diagnosis for any Substance Use Disorder (except nicotine or caffeine) in the 3 months prior to the screening visit.
8. Any medications (within 1 week of baseline or during the trial) that might confound the biomarker findings, including: Regular ingestion of NSAIDs or COX-2 inhibitors, or any use of oral steroids, immunosuppressants, interferon, chemotherapy (Patients will be instructed not to take an NSAID, COX-2 inhibitor or Aspirin in the 24 hours prior to a biomarker assessment visit).
9. Antibiotic treatment/consumption within four (4) weeks before baseline visit.
10. Patients who have taken foods or supplements with Probiotics later than two (2) weeks before baseline visit.
11. Active participation in other clinical studies with ongoing study visits.
12. Pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (interview version) | 8 weeks
  Decrease in depressive symtoms indicated by lower total score on mentioned scale, with 10 items, ranging from 0-60, a higher score indicating increased severity
"Inflammatory depressive symptoms" | 8 weeks
  Total composite score of the following items from the Patient Health Questionnaire (PHQ-9): item 3 (sleep problems), item 4 (lack of energy), and item 5 (appetite disturbance)

SECONDARY OUTCOMES:
Gastrointestinal Symptom Rating Scale for Irritable Bowel Syndrome (GSRS-IBS) | 8 weeks
  Total Composite score indicate severity of gastrointestinal symtoms, ranging from 0-78
Dimensional Anhedonia Rating Scale (DARS) | 8 weeks
  Total Composite score of 17 items, measuring different hedonic domains.
WHO Disability Assessment Schedule (WHODAS) | 8 weeks
  Total Composite score of 36 items, measuring Health and disability within 6 different domains, ranging from 0-144.
Generalized Anxiety Disorder-7 (GAD-7) | 8 weeks
  Total Composite score of 7 items, measuring anxiety symtoms, ranging from 0-21.
Insomnia Severity Index (ISI) | 8 weeks
  Total Composite score of 7 items, ranging from 0-28
Fatigue Severity Scale (FSS) | 8 weeks
  Total Composite score of 9 items, measuring severity of fatigue, ranging from 1-63
Wechsler Adult Intelligence Scale (WAIS-IV) | 8 weeks
  Two Composite scores of two tests measuring cognitive functioning. Symbol search, ranging from 0-60 and Digit symbol coding test ranging from 0-135.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lindqvist, PhD, Principal Investigator — Region Skane
Locations (1):
- Psychiatry Clinic, Lund, Region Skåne, Lund, Sweden

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT03660280/SAP_000.pdf